CLINICAL TRIAL: NCT00171132
Title: A 26-week Double-blind, Randomized, Multicenter Parallel-group Trial to Compare the Effects of Valsartan Versus Atenolol on Exercise Capacity in Hypertensive Overweight Postmenopausal Women With Impaired Exercise Tolerance
Brief Title: VALENCE: Valsartan Versus Atenolol on Exercise Capacity in Hypertensive Overweight Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489ADE21
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Postmenopausal; women; overweight; hypertension; impaired; exercise; capacity; valsartan; atenolol; hydrochlorothiazide
MeSH Terms: conditions — Hypertension; Overweight; Motor Activity | interventions — Valsartan; Atenolol; Hydrochlorothiazide

INTERVENTIONS:
Drug: valsartan
Drug: atenolol
Drug: hydrochlorothiazide

SUMMARY:
The purpose of the study is to show that valsartan compared to atenolol has favorable effects on exercise capacity, quality of life, diastolic function and elevated blood pressure in hypertensive postmenopausal overweight women with impaired exercise tolerance despite normal left ventricular ejection fraction (LVEF).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) must be ≥ 27 and < 35
* Symptoms of impaired exercise capacity (e.g. who report shortness of breath on exertion when questioned) reported at Visit 1 or patients who have a history of shortness of breath which improved under diuretic therapy
* LV ejection fraction must be > 45% measured by echocardiography at Visit 2.
* Impaired exercise capacity measured by VO2max at Visit 4:

VO2max >14 and < 22 ml ⋅kg-1 ⋅min-1

Exclusion Criteria:

* Mean sitting diastolic blood pressure (MSDBP) ≥ 110 mmHg and/or Mean sitting systolic blood pressure (MSSBP) ≥ 180 mmHg
* LVEF ≤ 45 %
* Inability to completely discontinue all previous antihypertensive medications safely for the duration of the study
* Heavy smokers (>20 cigarettes/day)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in exercise capacity measured by oxygen consumption during exercise testing, after 26 weeks

SECONDARY OUTCOMES:
Change from baseline in diastolic heart function after 26 weeks, measured by echocardiography
Change from baseline in heart rate and blood pressure,
during exercise testing after 26 weeks
Change from baseline in heart size after 26 weeks, measured by echocardiography
Change from baseline in quality of life measures after 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Dusing R, Handrock R, Klebs S, Tousset E, Vrijens B. Impact of supportive measures on drug adherence in patients with essential hypertension treated with valsartan: the randomized, open-label, parallel group study VALIDATE. J Hypertens. 2009 Apr;27(4):894-901. doi: 10.1097/HJH.0b013e328323f9be. PMID 19300114